CLINICAL TRIAL: NCT02802215
Title: Metformin for Prevention of Gestational Diabetes in Pregnant Women With Polycystic Ovarian Syndrome: Randomized Controlled Trial (RCT )
Brief Title: Metformin for Prevention Gestational Diabetes in Pregnant Women With Polycystic Ovarian Syndrome
Acronym: MGDPCOS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Assistant professor of Obstetric and Gynecology Faculty of medicine Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MGDPCOS
Record Dates: First submitted 2016-05-07; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2015-12

CONDITIONS: Polycystic Ovary Syndrome; Diabetes, Gestational
Keywords: Diabetes Mellitus; Pregnancy
MeSH Terms: conditions — Polycystic Ovary Syndrome; Diabetes, Gestational; Diabetes Mellitus | interventions — Metformin; Folic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin group (Active Comparator): 40 women will receive metformin in dose of 1500 mg per day orally (500 mg every 8 hrs in the middle of meal) starting from 12th week of gestation till delivery.
  Interventions: Drug: metformin
- control group (Placebo Comparator): 40 women will receive placebo which will be folic acid 500 micro gram which looks like metformin tablet.
  Interventions: Drug: placebo (folic acid )

INTERVENTIONS:
Drug: metformin — Metformin group will receive 1500 mg of metformin per day orally ( 500 mg every 8hrs in the middle of meal) starting from 12th week of gestation till delivery.
  Other Names: cidophage
  Arms: Metformin group
Drug: placebo (folic acid ) — 500 micro gram of folic acid every 8 hrs
  Other Names: folicap
  Arms: control group

SUMMARY:
Randomized, placebo controlled clinical trial that evaluate the role of taking metformin therapy during pregnancy in women with polycystic ovarian syndrome(PCOS) in reducing the development of gestational diabetes(GDM) and improving pregnancy outcomes.

DETAILED DESCRIPTION:
The study will include a total of 80 pregnant women who fulfill the inclusion and exclusion criteria. Participants will be distributed into two groups :

Group A: Active one (40 women) will receive metformin in a dose of 1500mg per day (500mg every 8hrs in the middle of meal), starting from 12th week of gestation till delivery.

Group B: control group (40 women) will receive placebo which will be folic acid 500 micro gram which looks like metformin tablet.

80 opaque envelope will be numbered serially from 1-80, in each envelope paper containing the group to which the participants will be allocated according to randomization table .The envelopes will be put in one box and when the first patient arrives the first envelope will be open and the patient will be allocated according to the paper inside.

Detection of glucose intolerance will be done using oral glucose tolerance test (OGTT), which based on 75 gm to exclude any case of pre-gestational DM. BMI and blood pressure will be also assessed for all cases at entry of the study.

Follow up of all cases in antenatal care clinic, with clinical assessment including weight gain, blood pressure, urine examination for proteinuria and fetal well being tests.

Detection of development of GDM or even glucose intolerance will be by using (OGTT), which based on 75 gm glucose between 24th-28th wk and also can be repeated between 32th- 34th wk of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* All women had confirmed diagnosis of PCOS before pregnancy according to revised 2003 Rotterdam criteria.
* Age more than 20 and more than 40 years.
* BMI ranging from (25_35 )
* Written and signed informed consent is given from the patient to participate in the study.

Exclusion Criteria:

* Women with pre-gestational diabetes mellitus confirmed by 2hrs OGTT.
* Patients who take metformin in the first 12 wk of pregnancy.
* Patients who are unwilling to participate in the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with gestational diabetes by measuring plasma glucose levels ( mg / dl ). | 24th -28th week gestation
  Diagnosis of GDM when these values are met or exceed fasting plasma glucose level (92 mg/dl).1hr level is (180 mg/dl) and 2hrs level is (153 mg/dl).

SECONDARY OUTCOMES:
Fetal adverse effects | from 12th week gestation till delivery
  Recorded in Case Record Form
Maternal adverse effects | from 12th week gestation till delivery
  Recorded in Case Record Form

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E elbohoty, MD, Principal Investigator — Ain Shams University; Reda k Mokhtar, MD, Principal Investigator — Ain Shams University; mai R ibrahim, MBBCH, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes